CLINICAL TRIAL: NCT04249687
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of QM1114-DP for the Treatment of Moderate to Severe Lateral Canthal Lines
Brief Title: Treatment of Moderate to Severe Lateral Canthal Lines
Acronym: READY-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43QM1901
Record Dates: First submitted 2020-01-07; First posted 2020-01-31 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2021-03

CONDITIONS: Lateral Canthal Lines
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): QM1114-DP, a Botulinum Toxin Type A (BoNT-A); Mode of administration: intramuscular injection
  Interventions: Biological: botulinum toxin
- Placebo (Placebo Comparator): A buffered solution; Mode of administration: intramuscular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: botulinum toxin — neuromodulator
  Other Names: QM1114-DP
  Arms: Treatment
Biological: Placebo — placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of a single dose of QM1114-DP compared to placebo for the treatment of moderate to severe LCL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Moderate to severe LCL at maximum smile as assessed by the Investigator.
3. Moderate to severe LCL at maximum smile as assessed by the subject.

Exclusion Criteria:

1. Previous use of any Botulinum toxin treatment in facial areas within 9 months prior to study treatment.
2. Female who is pregnant, breast feeding, or intends to conceive a child during the study.
3. Known allergy or hypersensitivity to any component of the investigational product (QM1114-DP) or any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Dermatology Cosmetic Laser Medical Associates, San Diego, California
  - Art of Skin, MD, Solana Beach, California
  - Siperstein Dermatology Group, PLLC, Boynton Beach, Florida
  - Facial Plastic Surgicenter, Ltd, Baltimore, Maryland
  - The Center for Dermatology, Cosmetic & Laser Surgery, Mount Kisco, New York
  - Rochester Dermatologic Surgery, Ltd, Victor, New York
  - Aesthetic Solutions, PA, Chapel Hill, North Carolina
- Canada (2):
  - Dr. Shannon Humphrey, Inc, Vancouver, British Columbia
  - Pacific Dermaesthetics, Inc, Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 230 | 73
Completed | 223 | 67
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 230 | 73 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (11.12) | 48.2 (11.48) | 50.1 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 63 | 263
  Male | 30 | 10 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 1 | 4
  White | 215 | 67 | 282
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥ 2-grade Improvement From Baseline on the Lateral Canthal Line Investigator and Subject Assessments at Maximum Smile at One Month.
Description: The investigator and subject evaluate the subject's LCL severity using a 4-grade scale (0 = none and 3 = severe)
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 204 | 69
Participants | 106 | 1
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects Who Achieve Grade 0 or 1 in Lateral Canthal Line Investigator Scale at Maximum Smile.
Time Frame: One Month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 200 | 68
Participants | 175 | 8
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/73
Serious Adverse Events (participants affected / at risk) | 3/230 | 1/73
Other Adverse Events (participants affected / at risk) | 20/230 | 12/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=230) | Placebo (N=73)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=230) | Placebo (N=73)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 11 (12) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04249687/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT04249687/SAP_001.pdf